CLINICAL TRIAL: NCT02211001
Title: Comparative Study of Strenght, Endurance, Flexibility of Muscle Trunk Between the Techniques: Global Postural Reeducation , Pilates and Segmented Dynamic Exercises.
Brief Title: Pilates, Postural Global Reeducation and Ball Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cintia Domingues de Freitas, Physical Therapist, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1159-8500
Record Dates: First submitted 2014-08-01; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Strength, Muscle; Endurance , Physical; Flexibility
Keywords: Exercise Movement Techniques; Exercise Therapy; Physical Therapy Modalities.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pilates Group (Experimental): The individuals were treated with Mat Pilates Method.
  Interventions: Other: Pilates Group
- Segmented Dynamic Exercises Group (Experimental): The individual were treated with ball exercises.
  Interventions: Other: Segmented Dynamic Exercises Group
- Global Postural Reeducation Group (Experimental): The individuals were treated with postures of Souchard Method.
  Interventions: Other: Global Postural Reeducation

INTERVENTIONS:
Other: Pilates Group — The exercises were applied once a week during eight weeks.
  Arms: Pilates Group
Other: Segmented Dynamic Exercises Group — The exercises were applied once a week during eight weeks. once a week for eight weeks.
  Arms: Segmented Dynamic Exercises Group
Other: Global Postural Reeducation — The exercises were applied once a week during eight weeks.
  Arms: Global Postural Reeducation Group

SUMMARY:
The purpose of this study is to evaluate and compare the effects of three Exercise Movement Techniques Global Postural Reeducation(RPG), Pilates method and Segmented Dynamic Exercises (SDE) regarding muscular strength and endurance of the trunk, spine mobility and flexibility of the posterior muscle chain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Healthy young adults who do not practice regular exercise
* The individuals could not have prior experience with the techniques covered in this study
* They could not report a history of pain,disease, neurological or orthopedic surgeries in column , upper or lower limbs, joint laxity, nor have history of injury and hamstring muscles in the lower limbs, neurological disorders, obesity, rheumatic disease, labyrinthitis, deformities of the lower limbs and spine
* Individuals could not make use of drugs that affected his balance and muscle strength
* To be framed the individual should also have restricted movement in the test distance of the third finger to the ground

Exclusion Criteria:

* Individuals with excessive absences (more than 20% of sessions) or those who missed and could not reset the session in the same week were excluded -Individuals who needed to undergo some surgery or any medical treatment during the duration of the study, or those who give up without completing the minimum time of the intervention

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Abdominal Muscle Endurance: Crunch test (repetitions per minute) | Baseline and week eight
  Control Group: Baseline 30,86 Week eight 31,24 SDE Group: Baseline 25,06 Week eight 32,00 Pilates Group: Baseline 25,29 Week eight 34,14 RPG Group: Baseline 30,61 Week eight 36,17
Extensors Muscle Endurance:Sorenson test (seconds) | Baseline and week eight
  Control Group: Baseline 69,43 Week eight 69,67 SDE Group: Baseline 72,65 Week eight 112,76 Pilates Group: Baseline 73,67 Week eight 74,43 RPG Group: Baseline 77,39 Week eight 119,48
Toe-touch test right/left | Baseline and week eight
  Control Group: Baseline 14,61/14,87 Week eight 14,89/14,91 SDE Group: Baseline 12,95/13,2 Week eight 10,12/10,32 Pilates Group: Baseline 13,81/13,93 Week eight 11,90/12,01 RPG Group : Baseline 17,63/18,15 Week eight: 9,11/9,22
Strength of trunk muscles:Peak Torque(Newton metre Nm) flexors and extensor muscles of spine measured in the isokinetic dynamometer BIODEX | Baseline and week eight
  Extension Control Group Baseline 206,1 week eight 236,9 SDE Group Baseline 213,5 week eight 239,3 Pilates Group Baseline 228,5 week eight 243,8 RPG Group Baseline 242,5 week eight 280,3
  Flexion Control Group Baseline 114,3 week eight 117,7 SDE Group Baseline 113,2 week eight 121,2 Pilates Group Baseline 109,3 week eight 118,5 RPG Group Baseline 127,2 week eight 138,1
Strength of trunk muscles:Muscle Work (Joules) of flexors and extensor muscles of spine measured in the isokinetic dynamometer BIODEX | Baseline and week eight
  Extension Control Group Baseline 847,9 week eight 958,6 SDE Group Baseline 893,5 week eight 985,4 Pilates Group Baseline 982,1 week eight 973,0 RPG Group Baseline 1053,1 week eight 1233,0
  Flexion
  Control Group Baseline 455,8 week eight 499,8 SDE Group Baseline 492,0 week eight 491,2 Pilates Group Baseline 472,0 week eight 498,9 RPG Group Baseline 558,7 week eight 581,9

CONTACTS AND LOCATIONS:
Overall Officials: Cintia de Freitas, student, Principal Investigator — FMUSP
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Kloubec JA. Pilates for improvement of muscle endurance, flexibility, balance, and posture. J Strength Cond Res. 2010 Mar;24(3):661-7. doi: 10.1519/JSC.0b013e3181c277a6. PMID 20145572
- [Result] Barr KP, Griggs M, Cadby T. Lumbar stabilization: a review of core concepts and current literature, part 2. Am J Phys Med Rehabil. 2007 Jan;86(1):72-80. doi: 10.1097/01.phm.0000250566.44629.a0. PMID 17304690
- [Result] Marshall PW, Murphy BA. Core stability exercises on and off a Swiss ball. Arch Phys Med Rehabil. 2005 Feb;86(2):242-9. doi: 10.1016/j.apmr.2004.05.004. PMID 15706550
- [Result] Carter JM, Beam WC, McMahan SG, Barr ML, Brown LE. The effects of stability ball training on spinal stability in sedentary individuals. J Strength Cond Res. 2006 May;20(2):429-35. doi: 10.1519/R-18125.1. PMID 16686575
- [Result] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Result] Vanti C, Generali A, Ferrari S, Nava T, Tosarelli D, Pillastrini P. [ General postural rehabilitation in musculoskeletal diseases: scientific evidence and clinical indications]. Reumatismo. 2007 Jul-Sep;59(3):192-201. Italian. PMID 17898878
- [Result] Oliveri M, Caltagirone C, Loriga R, Pompa MN, Versace V, Souchard P. Fast increase of motor cortical inhibition following postural changes in healthy subjects. Neurosci Lett. 2012 Nov 14;530(1):7-11. doi: 10.1016/j.neulet.2012.09.031. Epub 2012 Sep 28. PMID 23022506